CLINICAL TRIAL: NCT06900751
Title: A Phase 1 Study of NEU-627 to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect in Healthy Volunteers
Brief Title: A Study to Assess NEU-627 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuron23 Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-627-MS101
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEU-627 (Experimental): Part A: Single-ascending dose cohorts; Part B: Multiple-ascending dose cohort; Part C: Open-label, food effect evaluation; and Part D: Open-label, determination of cerebrospinal concentration
  Interventions: Drug: NEU-627
- Placebo (Experimental): Part A: Single-ascending dose cohorts; Part B: Multiple-ascending dose cohort
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NEU-627 — Investigational medicinal product
  Arms: NEU-627
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Phase 1, randomized, double-blind, placebo-controlled study of NEU-627 designed to evaluate safety, tolerability, pharmacokinetics, pharmacodynamics, and food effect.

DETAILED DESCRIPTION:
This is a Phase 1 study that will utilize a randomized, double-blind placebo controlled single ascending dose schema, a 10-day multiple ascending dose schema, and open-label schemas to study food effect and to determine cerebrospinal fluid concentration of NEU-627. The study will evaluate safety, tolerability, pharmacokinetics, pharmacodynamics, and food effect of NEU-627 in male and female healthy volunteers between 18 to 60 years old, inclusive.

ELIGIBILITY:
Inclusion criteria:

Participants are eligible to be included in the study only if all of the following criteria apply.

1. Male and female participants must be 18-60 years, inclusive, at the time of signing the informed consent;
2. Participants must be in good general health according to the judgment of the Investigator per local guidance;
3. Participants who have a body mass index (BMI) of 18-32 kg/m2 (inclusive);
4. When engaging in sex with a woman of child-bearing potential, both the male participant and his female partner must use highly effective contraception;
5. Legally and ethically capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply.

1. Clinically significant infection and/or dermatological, cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, neurological, or psychiatric disease which could interfere with, or the treatment for which might interfere with, the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the participant's risk if he/she were to participate in the study;
2. Any history of malignant disease in the last 5 years;
3. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions;
4. Use of or plans to use systemic immunosuppressive or immunomodulating medications during the study or within 3 months prior to the first study drug administration;
5. Current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications;
6. Positive screen for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody/antigen;
7. History of active, latent, or inadequately treated tuberculosis infection.

Additional details and criteria are outlined in the full study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of single and multiple doses of NEU-627 in healthy participants | Up to 10 days of dosing
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Evaluation of maximum concentration (Cmax) after single and multiple doses of NEU-627 | Up to 10 days of dosing
NEU-627 concentrations | Up to 10 days of dosing
Change from baseline of the corrected QT interval | Up to 10 days of dosing

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Grafton, Aukland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided